CLINICAL TRIAL: NCT00546663
Title: A Pilot Study to Evaluate the Tolerability of Inhaled 7% Hypertonic Saline in Infants With Cystic Fibrosis
Brief Title: Tolerability of Inhaled Hypertonic Saline in Infants With Cystic Fibrosis
Acronym: ISIS Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CF Therapeutics Development Network Coordinating Center (Network)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS001
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, hypertonic saline
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label (Experimental)
  Interventions: Drug: inhaled 7% hypertonic saline (HS)

INTERVENTIONS:
Drug: inhaled 7% hypertonic saline (HS) — 7% hypertonic saline administered twice daily for 14 days by nebulization.
  A Pari Sprint Junior nebulizer equipped with a Pari Baby face mask and a Pari Proneb compressor will be used to administer the HS (PARI Respiratory Equipment, Inc., Midlothian, VA).
  To minimize the risk of cough and bronchospasm with HS inhalation, infants will be pre-treated prior to each dose of HS with albuterol by metered dose inhaler
  Other Names: Hyper-Sal™, inhaled saline

SUMMARY:
This is an open-label pilot study of the safety and tolerability of 7% hypertonic saline inhaled twice daily for 14 days in infants with CF, 12 to 30 months of age.

DETAILED DESCRIPTION:
The efficacy and safety of hypertonic saline (HS) in CF patients over 6 years of age has been demonstrated in clinical trials of 2 to 48 weeks' duration. Based on these results, a large randomized, placebo-controlled trial of the efficacy and safety of 7% HS administered twice daily for 48 weeks to infants with CF, 4 to 15 months of age at enrollment, is planned (the Infant Study of Inhaled Saline (ISIS) trial). It is anticipated that 150 infants at up to 16 sites will be enrolled in the ISIS trial.

To date, the only evaluations of the safety of HS in infants with CF have been small single-dose studies. There has been no evaluation of the tolerability of chronic HS administration. The goal of this study is to assess the safety and tolerability of exposure to 14 days of 7% HS administered twice daily in infants with CF, prior to enrolling subjects in the planned large, randomized, controlled trial. Conduct of this study will provide evidence for the tolerability of chronic HS administration in infants with CF and estimates of the proportion of infants who do not tolerate chronic HS treatment. The results will be used to establish the appropriate measures of tolerability at enrollment in the ISIS trial, and to refine sample size estimates to account for withdrawal due to intolerance of HS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as defined by one or more clinical features of CF and a documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Informed consent by parent or legal guardian
* 12-30 months of age at enrollment

Exclusion Criteria:

* Wheezing at the baseline evaluation at the enrollment visit
* Oxygen saturation < 95 % at the baseline evaluation at the enrollment visit
* Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate, or new rhinorrhea, nasal congestion or rhinorrhea, with onset in the week preceding the enrollment visit
* Investigational drug use within 30 days prior to the enrollment visit
* Known intolerance of albuterol
* Current enrollment in a therapeutic clinical trial
* Condition or situation which, in the opinion of the investigator, would affect the ability of the patient or family to complete study procedures

Ages: 12 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The proportion of infants who are intolerant of single and repeated doses of HS according to protocol-defined criteria | At the enrollment visit, during the period of home administration (Days 0 to 14), and at the final study visit.

SECONDARY OUTCOMES:
New or increased cough, increased qualitative breathing rate, new or increased noisy breathing, or new or increased emesis at home as noted by parents on the daily symptom report | During the period of home administration (Days 0 to 14)
Change in respiratory rate, oxygen saturation, or cough frequency between the baseline measurement and measurements obtained after HS administration | At the enrollment visit
Change in respiratory rate, oxygen saturation, or cough frequency between the baseline value at the enrollment visit and the value at the final study visit | Over two weeks of study participation
Unanticipated adverse events | Over two weeks of study participation
Adherence, as measured by (1) the number of doses of HS administered per the home symptom report and (2) returned study drug vials | During the period of home administration (Days 0 to 14)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Rosenfeld, MD, MPH, Principal Investigator — Seattle Children's Hospital; Stephanie Davis, MD, Principal Investigator — University of North Carolina; Felix Ratjen, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada